CLINICAL TRIAL: NCT01061541
Title: A Phase II, Double-blind, Randomized Study to Compare the Immunogenicity, Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Tritanrix™-HepB/Hib2.5 to GSK Biologicals' Tritanrix™-HepB/Hiberix™ When Administered as a Three-dose Primary Vaccination Course to Healthy Infants at 6, 10 and 14 Weeks of Age. A Dose of Unconjugated Hib Vaccine (Plain PRP Booster) Will be Administered at the Age of 10 Months to 50% of the Subjects
Brief Title: Immunogenicity, Safety & Reactogenicity of GSK Vaccine Tritanrix™-HepB/Hib2.5 Compared to GSK Vaccine Tritanrix™-HepB/Hiberix™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208108/091; 208108/092 (Other: GSK)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b
Keywords: Pertussis; Tetanus; Hiberix™; Hepatitis B; DTPw-HBV vaccine; Tritanrix™-HepB; Haemophilus influenzae type b; Diphtheria; Hib vaccine
MeSH Terms: conditions — Haemophilus Infections; Whooping Cough; Tetanus; Hepatitis B; Diphtheria | interventions — Hiberix

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Tritanrix™-HepB low thio /; Biological: Hib 2.5; Biological: Unconjugated Hib vaccine (plain PRP)
- Group B (Active Comparator)
  Interventions: Biological: Tritanrix™-HepB; Biological: Hiberix™; Biological: Unconjugated Hib vaccine (plain PRP)

INTERVENTIONS:
Biological: Tritanrix™-HepB low thio / — One dose as intramuscular injection at 6, 10 and 14 weeks of age.
  Arms: Group A
Biological: Hib 2.5 — One dose as intramuscular injection at 6, 10 and 14 weeks of age.
  Arms: Group A
Biological: Tritanrix™-HepB — One dose as intramuscular injection at 6, 10 and 14 weeks of age.
  Arms: Group B
Biological: Hiberix™ — One dose as intramuscular injection at 6, 10 and 14 weeks of age.
  Arms: Group B
Biological: Unconjugated Hib vaccine (plain PRP) — One dose as intramuscular injection at 10 months of age

SUMMARY:
In order to reduce the amount of thiomersal in its vaccines, GSK Biologicals has developed a DTPw-HBV vaccine with low thiomersal content (Tritanrix™- HepB low thio). This vaccine is to be used in combination with a Hib low dose vaccine containing 2.5µg of PRP antigen (Hib 2.5). The purpose of this study is to generate clinical data with Tritanrix™-HepB low thio vaccine when extemporaneously mixed with Hib 2.5 vaccine. The control group will receive Tritanrix™-HepB/Hiberix™.

Subjects received primary vaccination in study 208108/091 (double blind). Of these subjects 50% were randomised to participate in the PRP challenge study (208108/092) (open), and all subjects will be invited to participate in a booster study DTPWHBV=HIB2.5-093 (101477).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 8 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks.
* Born to a mother proven seronegative for HBsAg.

Exclusion Criteria:

* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days before each dose of vaccine, with the exception of oral polio vaccine (OPV).
* Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B and/or Hib.
* History of, or intercurrent, diphtheria, tetanus, pertussis, hepatitis B and/or Hib disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or history.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Other conditions which in the opinion of the investigator may potentially interfere with interpretation of study outcomes.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2003-08; Primary Completion 2004-01 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
anti-PRP antibody concentration above a protocol defined cut-off value. | One month after the third dose of the primary vaccination course.

SECONDARY OUTCOMES:
anti-HBs antibody concentration | One month after the third dose of the primary vaccination course
anti-PRP antibody concentration | One month after the third dose of the primary vaccination course
anti-tetanus antibody concentration | One month after the third dose of the primary vaccination course
anti-diphtheria antibody concentration | One month after the third dose of the primary vaccination course
anti-Bordetella pertussis (BPT) antibody concentration | One month after the third dose of the primary vaccination course
Vaccine response to Bordetella pertussis antigen. | One month after the third dose of the primary vaccination course
Seropositivity/seroprotection rates and GMCs for antibodies against all vaccine antigens | Before the first dose of the primary vaccination course
anti-PRP antibody concentration | Before and one month after the plain PRP challenge dose.
Occurrence of solicited symptoms | During the 4-day follow-up period after each dose
Occurrence of unsolicited symptoms | During the 31-day follow-up period after each dose
Occurrence of serious adverse events | Over the full course of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Gatchalian SR, Ramakrishnan G, Bock HL, Lefevre I, Jacquet JM. Immunogenicity, reactogenicity and safety of three-dose primary and booster vaccination with combined diphtheria-tetanus-whole-cell pertussis-hepatitis B-reduced antigen content Haemophilus influenzae type b vaccine in Filipino children. Hum Vaccin. 2010 Aug;6(8):664-72. doi: 10.4161/hv.6.8.12155. PMID 20657177
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 208108/091 are summarised with study 208108/092 on the GSK Clinical Study Register.
- Available data/document: Statistical Analysis Plan: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208108/091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register